CLINICAL TRIAL: NCT07142902
Title: Gastroduodenal Full Thickness Resection Device Registry - gdFTRD® Registry
Status: Not yet recruiting | Type: Observational
Sponsor: Ovesco Endoscopy AG (Industry)
Collaborators: novineon CRO GmbH (Unknown)
Responsible Party: Sponsor
Other Study IDs: F-2024-112
Record Dates: First submitted 2025-07-25; First posted 2025-08-27 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2025-08

CONDITIONS: Subepithelial Gastrointestinal Tumors; Adenoma
Keywords: gdFTRD; gastroduodenal full thickness resection; endoscopic full thickness resection; EFTR
MeSH Terms: conditions — Adenoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- All patients of legal age with given informed consent to data processing: All patients of legal age in whom the gdFTRD was used for treatment independently from the registry
  Interventions: Other: Data processing only, treatment is not part of the registry

INTERVENTIONS:
Other: Data processing only, treatment is not part of the registry — Treatment with the gdFTRD is part of the clinical routine, the registry only comprises data processing after treatment.

SUMMARY:
Endoscopic full-thickness resection (EFTR) is a therapeutic option for the treatment of challenging lesions such as subepithelial tumors (SETs) and epithelial neoplasia extending deeper than the mucosa or associated with significant fibrosis. EFTR may offer a less invasive treatment alternative relative to surgical approaches in selected patients.

The gastroduodenal FTRD System (gdFTRD System) is an instrument for endoscopic full-thickness resection or deep partial wall resection and diagnostic tissue acquisition through removal of suitable lesions in the stomach and duodenum.

The prospectively generated data of the gdFTRD registry shall be used to evaluate the application of the gdFTRD in clinical routine, to verify the acceptability of already known risks and to identify unknown risks and complications.

DETAILED DESCRIPTION:
The gdFTRD registry is a registry on cases completed with the gdFTRD System. The gdFTRD System is used for full-thickness resection but the procedure is not part of the study. Only data processing is conducted within the study. For data processing, an EDC system is used.

There are no patient reported outcomes, only physician-entered data on baseline, intervention/procedure, complications/adverse events and follow-up visits.

Automatic plausibility checks have been programmed for quality assurance. Furthermore, warnings and hints will be given on predefined entries not allowed or to double-check values out of normal ranges. No source data verification is planned but data management will check the entries for completeness.

No coding according to MEDRA or similar systems is planned. As the procedure is not part of the study, every participating site must operate according to their own SOPs. The sponsor and CRO have SOPs in place for conducting a study. Furthermore, data protection requirements and all applicable regulations are followed.

The sample size was calculated based results of peer-reviewed publications on the gdFTRD System. As only continuous and categorial variables will be assessed, no separate statistical analysis plan is planned. In case the collected data allows for exploratory post hoc subgroup analysis further tests can be done according to the descriptions in the protocol. Missing data will not be included in the analysis and shall not be imputed.

ELIGIBILITY:
Inclusion criteria:

* All patients of legal age in whom the gdFTRD was used for treatment in the upper GI tract (stomach and duodenum) independently from the registry and
* who gave informed consent to data processing

Exclusion criteria:

* Patients aged under 18 years
* Patients in whom the colonic FTRD, diagnostic FTRD or non-device assisted EFTR was used for treatment
* Patients who did not give informed consent to data processing

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients of legal age in whom the gdFTRD was used for treatment independently from the registry.
Sampling Method: Non-Probability Sample
Enrollment: 306 (Estimated)
Dates: Start 2025-08 (Estimated); Primary Completion 2030-08 (Estimated); Study Completion 2030-08 (Estimated)

PRIMARY OUTCOMES:
Technical success | Directly post-procedure
  Technical success (i.e. target lesion reached and resected; macroscopically complete)

SECONDARY OUTCOMES:
Full thickness resection | Up to 14 days post-procedure
  Full-thickness resection (i.e. histologically confirmed full-thickness resection)
R0 resection | Up to 14 days post-procedure
  R0 resection (i.e. histologically complete lesion resection)
Rate of curative resection (in case of malignant tumors) | Up to 14 days post-procedure
  Rate of curative resection (in case of malignant tumors)

OTHER OUTCOMES:
Incidence of procedure-related adverse events (Safety) | Intra-procedural and directly post-procedure
  Total procedure-related adverse events
Incidence of surgery due to procedure-related adverse events (Safety) | up to 2 weeks post-procedure
  Surgery due to a procedure-related adverse event
Incidence of post-interventional complications (Safety) | up to 2 weeks post-procedure
  Post-interventional complications
Incidence of further procedure-related complications (Safety) | up to 3 years post-procedure
  Other procedure-related complications

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Wannhoff, PD Dr. med., Principal Investigator — RKH Kliniken Ludwigsburg-Bietigheim gGmbH
Locations (3):
- Germany (3):
  - Universitätsklinikum Freiburg - Klinik für Innere Medizin II, Freiburg im Breisgau, Germany
  - RKH Kliniken Ludwigsburg-Bietigheim gGmbH, Ludwigsburg, Germany
  - Robert-Bosch-Krankenhaus, Stuttgart, Germany

IPD SHARING:
Plan to Share IPD: No
Anonymized data will be used for publication of all participant data.

REFERENCES:
- [Background] Exposed versus nonexposed endoscopic full-thickness resection for duodenal subepithelial lesions: a tertiary care center experience (with videos) Nabi, Zaheer et al. iGIE, Volume 2, Issue 2, 154 - 160.e2
- [Background] Hajifathalian K, Ichkhanian Y, Dawod Q, Meining A, Schmidt A, Glaser N, Vosoughi K, Diehl DL, Grimm IS, James T, Templeton AW, Samarasena JB, Chehade NEH, Lee JG, Chang KJ, Mizrahi M, Barawi M, Irani S, Friedland S, Korc P, Aadam AA, Al-Haddad M, Kowalski TE, Smallfield G, Ginsberg GG, Fukami N, Lajin M, Kumta NA, Tang SJ, Naga Y, Amateau SK, Kasmin F, Goetz M, Seewald S, Kumbhari V, Ngamruengphong S, Mahdev S, Mukewar S, Sampath K, Carr-Locke DL, Khashab MA, Sharaiha RZ. Full-thickness resection device (FTRD) for treatment of upper gastrointestinal tract lesions: the first international experience. Endosc Int Open. 2020 Oct;8(10):E1291-E1301. doi: 10.1055/a-1216-1439. Epub 2020 Sep 22. PMID 33015330
- [Background] Wannhoff A, Nabi Z, Moons LMG, Haber G, Ge PS, Dertmann T, Deprez PH, Korcz W, Bouvette C, Mueller J, Tribonias G, Grande G, Kim JJ, Weich A, Heinrich H, Mollenkopf M, George J, Pioche M, Azzolini F, Kouladouros K, Boger P, Hayee B, Bilal M, Bastiaansen BAJ, Caca K; Upper GI FTRD Study Group. International, Multicenter Analysis of Endoscopic Full-Thickness Resection of Duodenal Neuroendocrine Tumors. Am J Gastroenterol. 2025 Dec 1;120(12):2800-2809. doi: 10.14309/ajg.0000000000003409. Epub 2025 Mar 13. PMID 40079474
- [Background] Meier B, Schmidt A, Glaser N, Meining A, Walter B, Wannhoff A, Riecken B, Caca K. Endoscopic full-thickness resection of gastric subepithelial tumors with the gFTRD-system: a prospective pilot study (RESET trial). Surg Endosc. 2020 Feb;34(2):853-860. doi: 10.1007/s00464-019-06839-2. Epub 2019 Jun 11. PMID 31187233